CLINICAL TRIAL: NCT02901639
Title: Influence of Immediate Postpartum Contraception Counseling on the Rate of Unintended Pregnancy in Primigravida: A Randomized Controlled Study
Brief Title: Postpartum Contraception Counseling on the Rate of Unintended Pregnancy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PPCC
Record Dates: First submitted 2016-09-10; First posted 2016-09-15 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Improving Quality of Life
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- counseling group (Experimental): will receive counseling about contraceptive methods using illustrations through postpartum interview with the study
  Interventions: Other: counseling
- NO counseling (No Intervention): will not receive any counseling about contraceptive methods

INTERVENTIONS:
Other: counseling
  Arms: counseling group

SUMMARY:
Unwanted pregnancies are not only the major cause of maternal mortality and morbidity but are also a great social and financial burden on societies and countries. According to World-health-organization statistics, there are an estimated 200 million pregnancies around the world each year, and a third of these, 75 million, are unwanted. Unintended pregnancy also is a major health problem in the United States of America. In the 2002 National Survey of Family Growth assessment, 1.22 million, or 31%, were reported as unintended. When abortions were included, unintended pregnancies increased to 2.65 million, or 49% of all pregnancies

ELIGIBILITY:
Inclusion Criteria:

1. Age: above 18 years
2. Primigravida
3. Women who will accept to participate in

Exclusion Criteria:

1. Women who are not intended to use contraception
2. Multiparous
3. Women who refuse to participate in the study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2018-08 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
The difference in the rate of unintended pregnancy in both groups | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided